CLINICAL TRIAL: NCT03227016
Title: Phase I/II Study in Patients With Small Cell Lung Cancer (SCLC) of Veliparib in Combination With Topotecan
Brief Title: Study in Patients With SCLC of Veliparib in Combination With Topotecan
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central European Society for Anticancer Drug Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-II-011
Record Dates: First submitted 2016-08-01; First posted 2017-07-24 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Small Cell Lung Cancer SCLC
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — veliparib; Poly(ADP-ribose) Polymerase Inhibitors; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination Topo/Veli (Experimental): Topotecan and Veliparib in increasing doses
  Interventions: Drug: veliparib; Drug: Topotecan

INTERVENTIONS:
Drug: veliparib — Topotecan at increasing doses (1x or 2x per day) will be administered in each cycle.
  Other Names: PARP inhibitor
Drug: Topotecan — Topotecan at dose 1.25 mg/m2 will be administered in each cycle.
  Other Names: Hycamtin

SUMMARY:
Phase I/II Study in Patients With Small Cell Lung Cancer (SCLC) of Veliparib in Combination With Topotecan

DETAILED DESCRIPTION:
For this study sensitive or refractory SCLC patients (refractory to prior chemotherapy defined as having experienced no response or a relapse within 90 days after the end of chemotherapy) will be eligible. In total, around 130 patients will be enrolled, around 30 evaluable patients in phase I and 100 patients in phase II.

The study will consist of two parts:

A preceding Phase I part will be performed to identify the Recommended Dose of veliparib to be administered in the Phase II part in combination with topotecan at the dose regimen of 1.25 mg/m2 (on days 1-5 of a 3 week cycle [d1-5q21d]). Each patient will be subjected to an initial cycle of topotecan monotherapy (1.25 mg/m2 on day 1-5 of a 3 week cycle); this run-in cycle shall prove topotecan tolerance of the candidates. Only patients who do not reveal any DLTs receive further treatment with combination therapy. In a dose-escalating 3+3 design the RD of veliparib for the subsequent Phase II part of the study will be defined during a maximum of 5 cycles combination therapy.

The Phase II part will follow upon completion of Phase I.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥ 18 years of age
* Subject with progressive or recurrent ED-SCLC after first line platinum-based therapy, which is either histologically or cytologically confirmed
* Performance status (PS) 0-2 ECOG
* Adequate bone marrow reserve
* Total bilirubin < 2 x upper limit of normal
* AST and ALT < 2.5 x upper limit of normal, or < 5 x upper limit of normal in case of liver metastases
* Serum creatinine < 2 x upper limit of normal or creatinine clearance > 50 ml/min

Exclusion Criteria:

* Other anti-cancer chemotherapy or radiotherapy
* Symptomatic motor or sensory neuro-toxicities CTCAE > Grade 2 or any other unresolved toxicities from prior systemic anti-cancer therapy or radiotherapy CTCAE > Grade 1
* Known hypersensitivity to topotecan or veliparib
* Brain or meningeal metastasis (unless they are asymptomatic and not requiring systemic corticosteroid therapy)
* Major surgery within 6 weeks prior to first treatment on study (subjects must have completely recovered from any previous surgery prior to first treatment on study).
* History of cardiac events within the past 3 months
* Uncontrolled severe hypertension
* Abdominal or tracheo-oesophageal fistula, gastrointestinal perforation, or intra-abdominal abscess
* Uncontrolled nausea / vomiting / diarrhea
* Previous malignancy (other than SCLC) in the last 3 years, except basal cell cancer of the skin, pre-invasive cancer of the cervix, T1a prostate carcinoma or superficial bladder tumor [Ta, Tis and T1] that was cured in the opinion of the investigator.
* History of organ allograft
* Active (acute or chronic) or uncontrolled infection of bacterial, mycotic or viral genesis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
adverse events | 6 months
  adverse events related to study drug(s) qualifying as Dose-Limiting Toxicities (DLT)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim von Pawel, MD, Study Chair — Askelios Klinik München Gauting
Locations (1):
- Klinik München Gauting, München Gauting, Germany